CLINICAL TRIAL: NCT07058792
Title: Impact of Medjool Date Consumption on Labor and Delivery Outcomes
Acronym: Yumi Dates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-059
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spontaneous Labor
Keywords: Medjool dates

STUDY DESIGN:
Intervention Model Description: One group will receive dates and one group will receive routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dates consumption group (Experimental): Subjects will eat dates in addition to routine care
  Interventions: Other: Medjool dates
- No dates group (No Intervention): Subjects will receive routine care only.

INTERVENTIONS:
Other: Medjool dates — Medjool dates are a dried fruit.
  Arms: Dates consumption group

SUMMARY:
The proposed Medjool date randomized trial will help inform clinical practice regarding the utility of Medjool date consumption for labor onset by comparing the incidence of spontaneous labor with the need for labor induction in patients who have been randomized to consume Medjool dates from 34 weeks gestation through the day after delivery day. The study will secondarily investigate the relationship between date consumption and other important labor and delivery outcomes such as length of labor, need for oxytocin, dose of oxytocin and quantitative blood loss at delivery. This study will also explore the association between Medjool date consumption, perinatal hemoglobin levels, and perinatal diet quality. Assessing dietary intake is an essential component of this study to better understand the relationship between medjool date consumption and pregnancy/labor outcomes by controlling for it as a potential confounding factor. Furthermore, assessing dietary intake will provide insight on the impact medjool date consumption has on overall maternal diet quality.

DETAILED DESCRIPTION:
The study is a randomized controlled trial evaluating labor outcomes for pregnant patients who begin Medjool date consumption during the 34th week of pregnancy versus those who do not consume dates prior to labor. We aim to assess whether Medjool date consumption impacts labor and delivery outcomes, specifically incidence of spontaneous labor compared with need for labor induction.

Patients will be screened and recruited at their routine prenatal appointment prior to 34 weeks. Eligible patients who desire participation after a discussion of the potential risks/benefits of participation will be consented and enrolled into this randomized control trial. They will randomized into either the Standard Care/No Dates group or the Dates group during this initial visit.

Patients randomized to the Dates group will be provided 42 pre-portioned bags of Medjool dates and instructed to eat 3 dates a day from 34 weeks of pregnancy until delivery as well as 3 dates on the day of delivery and 3 dates on the day after delivery. They will additionally have a point-of-care glucose check one hour consuming dates on the day of delivery. Patient will have daily surveys administered via REDCap to document their date intake prior to their delivery admission.

All patients in the study will also be completing food diaries through a 3-day electronic diet records for two time points during the study. The diet records will be electronic and collected using the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool. ASA24 is a validated, web-based dietary assessment tool developed by the National Cancer Institute for research purposes. The two time points for the diet records are 3 days prior to 34 weeks pregnancy and 3 days after 34 weeks of pregnancy. Patient will receive unique login information to complete the dietary records on the ASA24 website.

Data will be abstracted from the electronic medical record and stored in a password protected REDCap database only available to the study team. Dietary data will be collected through the National Cancer Institute's ASA24 research-based dietary assessment tool.

The researchers aim to recruit up to 250 patients at the study institution.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy less than 36weeks 0 days gestational age
* Age ≥18 years old
* Has decision-making capacity and able to provide informed consent for research participation
* Able to speak, read and understand English
* Planned delivery at a Cleveland Clinic Institution

Exclusion Criteria:

* Pre-existing medical co-morbidities including hypertension, kidney disease, autoimmune conditions, diabetes
* Comorbidities of pregnancy including hypertensive disorders of pregnancy and gestational diabetes
* Abnormal genetic (aneuploidy) screening or diagnostic testing
* Patients with pregnancies complicated by major fetal anomalies
* Multifetal gestation
* Delivery at an outside institution
* Incomplete delivery data
* Planned cesarean delivery
* Planned induction of labor prior to 41 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female participants
Enrollment: 250 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of spontaneous labor | 13 weeks
  This is a clinical diagnosis. Labor is defined as regular uterine contractions with cervical change. This will be documented in the medical record by the clinical provider.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Ehrenberg, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plans to make IPD public.